CLINICAL TRIAL: NCT01965470
Title: Botswana Combination Prevention Project: -Evaluation Protocol (Protocol #1): Research Design and Impact Evaluation -Closed Clinical Cohort Protocol (Protocol #3) Implementation, Monitoring and Evaluation of Combination HIV Prevention Interventions in Rural and Peri-Urban Communities in Botswana
Brief Title: Botswana Combination Prevention Project
Acronym: BCPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Botswana Ministry of Health (Other Government); Harvard School of Public Health (HSPH) (Other); Tebelopele Voluntary Counseling and Testing Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: CDC-CGH-6475
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Prevention (Experimental): * Scale-up of HTC services during 2 annual HTC campaigns, with a target of >90% of adults having documentation of their HIV-infected status or documentation of an HIV-negative test in the preceding 12 months.
  * Scale-up of universal ART for all HIV-infected adults, with a target of >93% of HIV positive adults receiving ART.
  * Scale-up of retention in care and adherence interventions, with a target of ensuring that >95% of HIV-infected adults are virally suppressed with HIV-1 RNA <400 copies per ML..
  * Scale-up of linkage to MC services, with a target of ensuring >60% of HIV-negative men are circumcised.
  * Rapid strengthening of PMTCT services, with a target of >90% of women initiated on indefinite ART (Option B+) during pregnancy remaining in care and on treatment at 12 months post-delivery.
  Interventions: Other: Combination Prevention
- Enhanced Care (Active Comparator): Enhanced Care Communities will receive guidance and improved technical support for quality management and data systems at all local clinics at which individuals receive HIV care and treatment.
  Interventions: Other: Enhanced Care

INTERVENTIONS:
Other: Combination Prevention
  Arms: Combination Prevention
Other: Enhanced Care
  Arms: Enhanced Care

SUMMARY:
The BCPP study is designed to test the hypothesis that implementing an enhanced combination prevention package which includes provision of ART to all participants, regardless of CD4 count or HIV disease severity, will impact the HIV/AIDS epidemic by significantly reducing population-level, cumulative HIV incidence in a defined geographic area over a period of 3 years and will be cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* Protocol #1 - Baseline Household Survey (BHS): Permanent or part-time study community resident in any of the 30 study communities; Botswana citizen or spouse of a Botswana citizen; able to provide informed consent if ≥18 years old, or able to provide assent to complement a guardian's permission, if a minor (aged 16 or 17).
* Protocol #3 - Expanded treatment cohort: HIV-infected persons in Combination Prevention communities who are not yet on ART and are able to provide informed consent if ≥18 years old, or able to provide assent to complement a guardian's permission, if a minor (aged 16 or 17).

Exclusion Criteria:

* Persons who do not meet inclusion criteria.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2013-10-30 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Population-level, cumulative HIV incidence | 3 years
  Population-level cumulative HIV incidence will be measured in a cohort of HIV-negative persons identified from a 20% sample of eligible households in the 30 study communities followed annually.

SECONDARY OUTCOMES:
2. Population-level uptake of HIV testing and counseling (HTC), ART, VL Suppression, male circumcision (MC), and PMTCT services | 3 years
  Population-level uptake of each intervention will be measured in an annual survey of the 20% sample of eligible households in the 30 study communities and through analysis of routine program monitoring data.
Cost per additional infection averted | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Janet S Moore, PhD, Principal Investigator — Centers for Disease Control and Prevention; Myron Essex, DVM, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Refeletswe Lebelonyane, MD, Principal Investigator — Botswana Ministry of Health; Shenaaz El Halabi, MPH, Principal Investigator — Botswana Ministry of Health; Joseph Makhema, MBChB, FRCP, Principal Investigator — Botswana Harvard AIDS Institute Partnership; Shahin Lockman, MD, MS, Principal Investigator — Harvard School of Public Health (HSPH); Eric Tchetgen Tchetgen, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Molly Pretorius Holme, MS, Principal Investigator — Harvard School of Public Health (HSPH); Pam Bachanas, PhD, Principal Investigator — Centers for Disease Control and Prevention; Tafireyi Marukutira, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Botswana communities and Botswana Ministry of Health clinics, Multiple Locations, Multiple, Botswana

REFERENCES:
- [Background] Moyo S, Gaseitsiwe S, Mohammed T, Pretorius Holme M, Wang R, Kotokwe KP, Boleo C, Mupfumi L, Yankinda EK, Chakalisa U, van Widenfelt E, Gaolathe T, Mmalane MO, Dryden-Peterson S, Mine M, Lebelonyane R, Bennett K, Leidner J, Wirth KE, Tchetgen Tchetgen E, Powis K, Moore J, Clarke WA, Lockman S, Makhema JM, Essex M, Novitsky V. Cross-sectional estimates revealed high HIV incidence in Botswana rural communities in the era of successful ART scale-up in 2013-2015. PLoS One. 2018 Oct 24;13(10):e0204840. doi: 10.1371/journal.pone.0204840. eCollection 2018. PMID 30356287
- [Background] Novitsky V, Gaolathe T, Mmalane M, Moyo S, Chakalisa U, Yankinda EK, Marukutira T, Holme MP, Sekoto T, Gaseitsiwe S, Musonda R, van Widenfelt E, Powis KM, Khan N, Dryden-Peterson S, Bennett K, Wirth KE, Tchetgen ET, Bachanas P, Mills LA, Lebelonyane R, El-Halabi S, Makhema J, Lockman S, Essex M. Lack of Virological Suppression Among Young HIV-Positive Adults in Botswana. J Acquir Immune Defic Syndr. 2018 Aug 15;78(5):557-565. doi: 10.1097/QAI.0000000000001715. PMID 29771781
- [Background] Moyo S, Gaseitsiwe S, Powis KM, Pretorius Holme M, Mohammed T, Zahralban-Steele M, Yankinde EK, Maphorisa C, Abrams W, Lebelonyane R, Manyake K, Sekoto T, Mmalane M, Gaolathe T, Wirth KE, Makhema J, Lockman S, Clarke W, Essex M, Novitsky V. Undisclosed antiretroviral drug use in Botswana: implication for national estimates. AIDS. 2018 Jul 17;32(11):1543-1546. doi: 10.1097/QAD.0000000000001862. PMID 29762166
- [Background] Novitsky V, Prague M, Moyo S, Gaolathe T, Mmalane M, Yankinda EK, Chakalisa U, Lebelonyane R, Khan N, Powis KM, Widenfelt E, Gaseitsiwe S, Dryden-Peterson SL, Holme MP, De Gruttola V, Bachanas P, Makhema J, Lockman S, Essex M. High HIV-1 RNA Among Newly Diagnosed People in Botswana. AIDS Res Hum Retroviruses. 2018 Mar;34(3):300-306. doi: 10.1089/AID.2017.0214. Epub 2018 Jan 17. PMID 29214845
- [Background] Moyo S, Mohammed T, Wirth KE, Prague M, Bennett K, Holme MP, Mupfumi L, Sebogodi P, Moraka NO, Boleo C, Maphorisa CN, Seraise B, Gaseitsiwe S, Musonda RM, van Widenfelt E, Powis KM, Gaolathe T, Tchetgen Tchetgen EJ, Makhema JM, Essex M, Lockman S, Novitsky V. Point-of-Care Cepheid Xpert HIV-1 Viral Load Test in Rural African Communities Is Feasible and Reliable. J Clin Microbiol. 2016 Dec;54(12):3050-3055. doi: 10.1128/JCM.01594-16. Epub 2016 Oct 12. PMID 27733636
- [Background] Gaolathe T, Wirth KE, Holme MP, Makhema J, Moyo S, Chakalisa U, Yankinda EK, Lei Q, Mmalane M, Novitsky V, Okui L, van Widenfelt E, Powis KM, Khan N, Bennett K, Bussmann H, Dryden-Peterson S, Lebelonyane R, El-Halabi S, Mills LA, Marukutira T, Wang R, Tchetgen EJ, DeGruttola V, Essex M, Lockman S; Botswana Combination Prevention Project study team. Botswana's progress toward achieving the 2020 UNAIDS 90-90-90 antiretroviral therapy and virological suppression goals: a population-based survey. Lancet HIV. 2016 May;3(5):e221-30. doi: 10.1016/S2352-3018(16)00037-0. Epub 2016 Mar 24. PMID 27126489
- [Background] Novitsky V, Zahralban-Steele M, McLane MF, Moyo S, van Widenfelt E, Gaseitsiwe S, Makhema J, Essex M. Correction for Novitsky et al., Long-Range HIV Genotyping Using Viral RNA and Proviral DNA for Analysis of HIV Drug Resistance and HIV Clustering. J Clin Microbiol. 2016 Apr;54(4):1175. doi: 10.1128/JCM.00190-16. No abstract available. PMID 27016593
- [Background] Perriat D, Balzer L, Hayes R, Lockman S, Walsh F, Ayles H, Floyd S, Havlir D, Kamya M, Lebelonyane R, Mills LA, Okello V, Petersen M, Pillay D, Sabapathy K, Wirth K, Orne-Gliemann J, Dabis F; Universal Test and Treat Trials Consortium (UT3C). Comparative assessment of five trials of universal HIV testing and treatment in sub-Saharan Africa. J Int AIDS Soc. 2018 Jan;21(1):e25048. doi: 10.1002/jia2.25048. PMID 29314658
- [Background] Novitsky V, Zahralban-Steele M, Moyo S, Nkhisang T, Maruapula D, McLane MF, Leidner J, Bennett K; PANGEA Consortium; Wirth KE, Gaolathe T, Kadima E, Chakalisa U, Pretorius Holme M, Lockman S, Mmalane M, Makhema J, Gaseitsiwe S, DeGruttola V, Essex M. Mapping of HIV-1C Transmission Networks Reveals Extensive Spread of Viral Lineages Across Villages in Botswana Treatment-as-Prevention Trial. J Infect Dis. 2020 Nov 15;222(10):1670-1680. doi: 10.1093/infdis/jiaa276. Epub 2020 Jun 3. PMID 32492145
- [Background] Lebelonyane R, Mills LA, Mogorosi C, Ussery F, Marukutira T, Theu J, Kapanda M, Matambo S, Block L, Raizes E, Makhema J, Lockman S, Bachanas P, Moore J, Jarvis JN. Advanced HIV disease in the Botswana combination prevention project: prevalence, risk factors, and outcomes. AIDS. 2020 Dec 1;34(15):2223-2230. doi: 10.1097/QAD.0000000000002627. PMID 32694412
- [Background] Lockman S, Holme MP, Makhema J, Bachanas P, Moore J, Wirth KE, Lebelonyane R, Essex M. Implementation of Universal HIV Testing and Treatment to Reduce HIV Incidence in Botswana: the Ya Tsie Study. Curr HIV/AIDS Rep. 2020 Oct;17(5):478-486. doi: 10.1007/s11904-020-00523-0. PMID 32797382
- [Background] Lebelonyane R, Bachanas P, Block L, Ussery F, Abrams W, Roland M, Theu J, Kapanda M, Matambo S, Lockman S, Gaolathe T, Makhema J, Moore J, Jarvis JN. Rapid antiretroviral therapy initiation in the Botswana Combination Prevention Project: a quasi-experimental before and after study. Lancet HIV. 2020 Aug;7(8):e545-e553. doi: 10.1016/S2352-3018(20)30187-9. PMID 32763218
- [Background] Alwano MG, Bachanas P, Block L, Roland M, Sento B, Behel S, Lebelonyane R, Wirth K, Ussery F, Bapati W, Motswere-Chirwa C, Abrams W, Ussery G, Miller JA, Bile E, Fonjungo P, Kgwadu A, Holme MP, Del Castillo L, Gaolathe T, Leme K, Majingo N, Lockman S, Makhema J, Bock N, Moore J. Increasing knowledge of HIV status in a country with high HIV testing coverage: Results from the Botswana Combination Prevention Project. PLoS One. 2019 Nov 25;14(11):e0225076. doi: 10.1371/journal.pone.0225076. eCollection 2019. PMID 31765394
- [Background] Kebaabetswe P, Manyake K, Kadima E, Auletta-Young C, Chakalisa U, Sekoto T, Dintwa OM, Mmalane M, Makhema J, Lebelonyane R, Bachanas P, Plank R, Gaolathe T, Lockman S, Holme MP. Barriers and facilitators to linkage to care and ART initiation in the setting of high ART coverage in Botswana. AIDS Care. 2020 Jun;32(6):722-728. doi: 10.1080/09540121.2019.1640843. Epub 2019 Jul 12. PMID 31298037
- [Background] Chakalisa U, Wirth K, Bennett K, Kadima E, Manyake K, Gaolathe T, Bachanas P, Marukutira T, Lebelonyane R, Dryden-Peterson S, Butler L, Mmalane M, Makhema J, Roland ME, Pretorius-Holme M, Essex M, Lockman S, Powis KM. Self-reported risky sexual practices among adolescents and young adults in Botswana. South Afr J HIV Med. 2019 Jun 26;20(1):899. doi: 10.4102/sajhivmed.v20i1.899. eCollection 2019. PMID 31308965
- [Background] Moyo S, Gaseitsiwe S, Zahralban-Steele M, Maruapula D, Nkhisang T, Mokaleng B, Mohammed T, Ditlhako TR, Bareng OT, Mokgethi TP, van Widenfelt E, Pretorius-Holme M, Mine MO, Raizes E, Yankinda EK, Wirth KE, Gaolathe T, Makhema JM, Lockman S, Essex M, Novitsky V. Low rates of nucleoside reverse transcriptase inhibitor and nonnucleoside reverse transcriptase inhibitor drug resistance in Botswana. AIDS. 2019 May 1;33(6):1073-1082. doi: 10.1097/QAD.0000000000002166. PMID 30946161
- [Background] Lasry A, Bachanas P, Suraratdecha C, Alwano MG, Behel S, Pals S, Block L, Moore J. Cost of Community-Based HIV Testing Activities to Reach Saturation in Botswana. AIDS Behav. 2019 Apr;23(4):875-882. doi: 10.1007/s10461-019-02408-9. PMID 30673897
- [Background] Molebatsi K, Gabaitiri L, Mokgatlhe L, Moyo S, Gaseitsiwe S, Wirth KE, DeGruttola V, Tchetgen Tchetgen E. Efficient estimation of human immunodeficiency virus incidence rate using a pooled cross-sectional cohort study design. Stat Med. 2020 Oct 30;39(24):3255-3271. doi: 10.1002/sim.8661. Epub 2020 Sep 1. PMID 32875624
- [Background] Bareng OT, Seselamarumo S, Seatla KK, Choga WT, Bakae B, Maruapula D, Kelentse N, Moraka NO, Mokaleng B, Mokgethi PT, Ditlhako TR, Pretorius-Holme M, Mbulawa MB, Lebelonyane R, Bile EC, Gaolathe T, Shapiro R, Makhema JM, Lockman S, Essex M, Novitsky V, Mpoloka SW, Moyo S, Gaseitsiwe S. Doravirine-associated resistance mutations in antiretroviral therapy naive and experienced adults with HIV-1 subtype C infection in Botswana. J Glob Antimicrob Resist. 2022 Dec;31:128-134. doi: 10.1016/j.jgar.2022.08.008. Epub 2022 Aug 13. PMID 35973671
- [Background] Bhebhe L, Moyo S, Gaseitsiwe S, Pretorius-Holme M, Yankinda EK, Manyake K, Kgathi C, Mmalane M, Lebelonyane R, Gaolathe T, Bachanas P, Ussery F, Letebele M, Makhema J, Wirth KE, Lockman S, Essex M, Novitsky V, Ragonnet-Cronin M. Epidemiological and viral characteristics of undiagnosed HIV infections in Botswana. BMC Infect Dis. 2022 Aug 28;22(1):710. doi: 10.1186/s12879-022-07698-4. PMID 36031617
- [Background] Marukutira T, Ussery F, Kadima E, Mills LA, Moore J, Block L, Bachanas P, Davis S, Schissler T, Mosha R, Komotere O, Diswai T, Ntsuape C, Lebelonyane R, Bock N. Male circumcision uptake during the Botswana Combination Prevention Project. PLoS One. 2022 Jun 15;17(6):e0269178. doi: 10.1371/journal.pone.0269178. eCollection 2022. PMID 35704556
- [Background] Ussery F, Bachanas P, Alwano MG, Lebelonyane R, Block L, Wirth K, Ussery G, Sento B, Gaolathe T, Kadima E, Abrams W, Segolodi T, Hader S, Lockman S, Moore J. HIV Incidence in Botswana Rural Communities With High Antiretroviral Treatment Coverage: Results From the Botswana Combination Prevention Project, 2013-2017. J Acquir Immune Defic Syndr. 2022 Sep 1;91(1):9-16. doi: 10.1097/QAI.0000000000003017. PMID 35537094
- [Background] Bareng OT, Moyo S, Zahralban-Steele M, Maruapula D, Ditlhako T, Mokaleng B, Mokgethi P, Choga WT, Moraka NO, Pretorius-Holme M, Mine MO, Raizes E, Molebatsi K, Motswaledi MS, Gobe I, Mohammed T, Gaolathe T, Shapiro R, Mmalane M, Makhema JM, Lockman S, Essex M, Novitsky V, Gaseitsiwe S. HIV-1 drug resistance mutations among individuals with low-level viraemia while taking combination ART in Botswana. J Antimicrob Chemother. 2022 Apr 27;77(5):1385-1395. doi: 10.1093/jac/dkac056. PMID 35229102
- [Background] Magosi LE, Zhang Y, Golubchik T, DeGruttola V, Tchetgen Tchetgen E, Novitsky V, Moore J, Bachanas P, Segolodi T, Lebelonyane R, Pretorius Holme M, Moyo S, Makhema J, Lockman S, Fraser C, Essex MM, Lipsitch M; Botswana Combination Prevention Project and PANGEA consortium. Deep-sequence phylogenetics to quantify patterns of HIV transmission in the context of a universal testing and treatment trial - BCPP/Ya Tsie trial. Elife. 2022 Mar 1;11:e72657. doi: 10.7554/eLife.72657. PMID 35229714
- [Background] Seatla KK, Maruapula D, Choga WT, Morerinyane O, Lockman S, Novitsky V, Kasvosve I, Moyo S, Gaseitsiwe S. Limited HIV-1 Subtype C nef 3'PPT Variation in Combination Antiretroviral Therapy Naive and Experienced People Living with HIV in Botswana. Pathogens. 2021 Aug 13;10(8):1027. doi: 10.3390/pathogens10081027. PMID 34451492
- [Derived] Kelepile M, Kebotsamang K, Mawi M, Molebatsi K, Molefe-Baikai OJ, Babayani N, Grady SC, Mogaetsho GE, Moshomo T, Kgotlaetsile K, Leeme T, Gaolathe T, Mosepele M. Spatial distribution of central obesity in rural and peri urban communities of Botswana: a nested Botswana Combination Prevention Project (BCPP) cross-sectional study. BMC Public Health. 2026 Jan 26. doi: 10.1186/s12889-026-26247-1. Online ahead of print. PMID 41588385
- [Derived] Moshomo T, Mawi M, Williams CG, Molebatsi K, Masupe T, Manyake K, Lockman S, Molefe-Baikai OJ, Leero A, Jarvis JN, Gaolathe T, Mosepele M. Comparison of central obesity prevalence among adults living with and without HIV in Botswana: a cross-sectional study. BMJ Open. 2025 Apr 21;15(4):e096170. doi: 10.1136/bmjopen-2024-096170. PMID 40258642
- [Derived] Cui Y, Moyo S, Pretorius Holme M, Hurwitz KE, Choga W, Bennett K, Chakalisa U, San JE, Manyake K, Kgathi C, Diphoko A, Gaseitsiwe S, Gaolathe T, Essex M, Tchetgen Tchetgen E, Makhema JM, Lockman S. Predictors of HIV seroconversion in Botswana. AIDS. 2025 Mar 1;39(3):290-297. doi: 10.1097/QAD.0000000000004055. Epub 2024 Nov 4. PMID 39497537
- [Derived] Zuze BJL, Radibe BT, Choga WT, Bareng OT, Moraka NO, Maruapula D, Seru K, Mokgethi P, Mokaleng B, Ndlovu N, Kelentse N, Pretorius-Holme M, Shapiro R, Lockman S, Makhema J, Novitsky V, Seatla KK, Moyo S, Gaseitsiwe S. Fostemsavir resistance-associated polymorphisms in HIV-1 subtype C in a large cohort of treatment-naive and treatment-experienced individuals in Botswana. Microbiol Spectr. 2023 Dec 12;11(6):e0125123. doi: 10.1128/spectrum.01251-23. Epub 2023 Oct 12. PMID 37823653
- [Derived] Kotokwe K, Moyo S, Zahralban-Steele M, Holme MP, Melamu P, Koofhethile CK, Choga WT, Mohammed T, Nkhisang T, Mokaleng B, Maruapula D, Ditlhako T, Bareng O, Mokgethi P, Boleo C, Makhema J, Lockman S, Essex M, Ragonnet-Cronin M, Novitsky V, Gaseitsiwe S, Pangea Consortium. Prediction of Coreceptor Tropism in HIV-1 Subtype C in Botswana. Viruses. 2023 Jan 31;15(2):403. doi: 10.3390/v15020403. PMID 36851617
- [Derived] Resch SC, Foote JHA, Wirth KE, Lasry A, Scott JA, Moore J, Shebl FM, Gaolathe T, Feser MK, Lebelonyane R, Hyle EP, Mmalane MO, Bachanas P, Yu L, Makhema JM, Holme MP, Essex M, Alwano MG, Lockman S, Freedberg KA. Health Impact and Cost-Effectiveness of HIV Testing, Linkage, and Early Antiretroviral Treatment in the Botswana Combination Prevention Project. J Acquir Immune Defic Syndr. 2022 Aug 1;90(4):399-407. doi: 10.1097/QAI.0000000000002996. Epub 2022 Apr 14. PMID 35420554
- [Derived] Lebelonyane R, Bachanas P, Block L, Ussery F, Alwano MG, Marukutira T, El Halabi S, Roland M, Abrams W, Ussery G, Miller JA, Lockman S, Gaolathe T, Holme MP, Hader S, Mills LA, Wirth K, Bock N, Moore J. To achieve 95-95-95 targets we must reach men and youth: High level of knowledge of HIV status, ART coverage, and viral suppression in the Botswana Combination Prevention Project through universal test and treat approach. PLoS One. 2021 Aug 10;16(8):e0255227. doi: 10.1371/journal.pone.0255227. eCollection 2021. PMID 34375343
- [Derived] Bachanas P, Alwano MG, Lebelonyane R, Block L, Behel S, Raizes E, Ussery G, Wang H, Ussery F, Pretorius Holme M, Sexton C, Pals S, Lasry A, Del Castillo L, Hader S, Lockman S, Bock N, Moore J. Finding, treating and retaining persons with HIV in a high HIV prevalence and high treatment coverage country: Results from the Botswana Combination Prevention Project. PLoS One. 2021 Apr 21;16(4):e0250211. doi: 10.1371/journal.pone.0250211. eCollection 2021. PMID 33882092
- [Derived] Wirth KE, Gaolathe T, Pretorius Holme M, Mmalane M, Kadima E, Chakalisa U, Manyake K, Matildah Mbikiwa A, Simon SV, Letlhogile R, Mukokomani K, van Widenfelt E, Moyo S, Bennett K, Leidner J, Powis KM, Lebelonyane R, Alwano MG, Jarvis J, Dryden-Peterson SL, Kgathi C, Moore J, Bachanas P, Raizes E, Abrams W, Block L, Sento B, Novitsky V, El-Halabi S, Marukutira T, Mills LA, Sexton C, Pals S, Shapiro RL, Wang R, Lei Q, DeGruttola V, Makhema J, Essex M, Lockman S, Tchetgen Tchetgen EJ. Population uptake of HIV testing, treatment, viral suppression, and male circumcision following a community-based intervention in Botswana (Ya Tsie/BCPP): a cluster-randomised trial. Lancet HIV. 2020 Jun;7(6):e422-e433. doi: 10.1016/S2352-3018(20)30103-X. PMID 32504575
- [Derived] Marukutira T, Block L, Alwano MG, Behel S, Jarvis JN, Chakalisa U, Powis K, Novitsky V, Bapati W, Wang H, Ussery F, Lebelonyane R, Mills LA, Moore J, Bachanas P. Comparison of knowledge of HIV status and treatment coverage between non-citizens and citizens: Botswana Combination Prevention Project (BCPP). PLoS One. 2019 Aug 29;14(8):e0221629. doi: 10.1371/journal.pone.0221629. eCollection 2019. PMID 31465494
- [Derived] Makhema J, Wirth KE, Pretorius Holme M, Gaolathe T, Mmalane M, Kadima E, Chakalisa U, Bennett K, Leidner J, Manyake K, Mbikiwa AM, Simon SV, Letlhogile R, Mukokomani K, van Widenfelt E, Moyo S, Lebelonyane R, Alwano MG, Powis KM, Dryden-Peterson SL, Kgathi C, Novitsky V, Moore J, Bachanas P, Abrams W, Block L, El-Halabi S, Marukutira T, Mills LA, Sexton C, Raizes E, Gaseitsiwe S, Bussmann H, Okui L, John O, Shapiro RL, Pals S, Michael H, Roland M, DeGruttola V, Lei Q, Wang R, Tchetgen Tchetgen E, Essex M, Lockman S. Universal Testing, Expanded Treatment, and Incidence of HIV Infection in Botswana. N Engl J Med. 2019 Jul 18;381(3):230-242. doi: 10.1056/NEJMoa1812281. PMID 31314967

DOCUMENTS (1):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT01965470/Prot_001.pdf